CLINICAL TRIAL: NCT04263831
Title: Low Dose IL-2 for the Treatment of Crohn's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Scott B. Snapper, MD PHD, Chief, Gastroenterology, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00032653; R01DK126448 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease
Keywords: Inflammatory bowel disease; Interleukin 2; Regulatory T Cells
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interleukin-2 (Experimental): Study drug: Interleukin-2 (aldesleukin, Proleukin, IL-2).
  Each subject will receive an 8-week course of once-daily, subcutaneously administered IL-2. There will be two dose cohorts. Each subject will be recruited into a single dose cohort and receive a single dose level of IL-2 throughout the study.
  The dose levels will be as follows:
  Cohort 1: 1.0x10^6 IU/m^2/day. Cohort 2: 1.25x10^6 IU/m^2/day.
  Interventions: Drug: Interleukin-2 (aldesleukin).

INTERVENTIONS:
Drug: Interleukin-2 (aldesleukin). — Description of intervention is covered in "Arm", above.

SUMMARY:
The purpose of this study is to determine the safety and maximum effective dose (MED) of Interleukin-2 in subjects with moderate-to-severe crohn's disease.

DETAILED DESCRIPTION:
Despite recent advances in treatment, a significant proportion of patients with Crohn's disease have suboptimal responses to medical therapy, leaving an urgent need to identify new therapies. One promising new approach to treat IBD is through the manipulation of regulatory T cells (Tregs). Tregs are an immune modulating subset of CD4+ lymphocytes that antagonize the activation and effector function of multiple immune cell types and promote tolerance to self-antigens. Adoptively transferred Tregs are effective in murine models of IBD. An alternative approach to disease management through Treg manipulation is to increase Treg numbers in vivo. Interleukin-2 (IL-2, Proleukin®) is a T cell growth factor. IL-2 is currently licensed for the treatment of metastatic renal cell carcinoma and metastatic melanoma. At low doses, IL-2 promotes the selective activation and expansion of Tregs in humans. Tregs constitutively express CD25, a component of the high-affinity IL-2R, while CD25 is only transiently expressed by activated conventional T effector cells. Low-dose (LD) IL-2 selectively expands Tregs in humans and is safe in chronic GvHD and other phase 1 and 2 clinical trials.

This is a phase 1b/2a clinical trial to assess the safety and the efficacy of LD SC IL-2 for the treatment of CD utilizing daily sc LD IL-2 for 8 weeks in CD patients to determine the maximum effective dose (MED) and safety profile, and to assess a signal of efficacy. We aim to determine in CD patients whether sc LD IL-2 modulates peripheral blood and lamina propria Tregs in vivo and correlates with clinical outcome. We will perform deep immunophenotyping in CD patients treated with LD IL-2 and comprehensively assess the effects of LD IL-2 on CD4+ Tregs and other immune cells in both peripheral and mucosal compartments, and correlate changes in immune phenotype with clinical outcome. Overall this trial is designed to determine the MED and safety profile of LD IL-2 in CD, to obtain a signal of efficacy, and to assess mechanistic underpinnings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-80 years. Maximum age limit for subjects recruited at BCH will be 30 years.
2. A diagnosis of CD made by standard clinical, radiological, endoscopic and histological criteria.

   a. A subset of patients with Ileostomies or colostomies will be permitted.
3. Adult subjects with moderate-to-severe CD (CDAI score 220-450)

   a. a modified CDAI will be used to assess patients with ileostomies/colostomies. Number of liquid stools per day will be substituted for number of bag empties per day.
4. Evidence of endoscopic inflammation accessible via ileocolonoscopy or ileoscopy

   1. Simple Endoscopic Score for CD (SES-CD) ≥ 6 or ≥ 4 for isolated ileal disease
   2. patients with ileostomies will be assessed as patients with isolated ileal disease via SES-CD.
5. Failure to tolerate or failure to respond to at least one conventional therapy with the intention of inducing or maintaining remission (including but not limited to oral corticosteroids, oral 5-aminosalicylates, azathioprine and/or 6-mercaptopurine, TNF alpha antagonist, anti-integrins, ustekinumab). Corticosteroid dependency (inability to taper oral corticosteroids without a recurrence of disease activity) is also included in this category.
6. Stable doses of concomitant medications, as defined in Section 5
7. A negative pregnancy test within 2 weeks prior to anticipated commencement of the study drug, in female subjects of child-bearing age. Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
8. The ability of adult participants who are able to make their own healthcare decisions to provide informed consent or the ability of a legal guardian to provide consent if the participant is a child (less than 18 years of age) or has mild intellectual disability and cannot consent for him or herself. In the event that a legal guardian provides consent, the study participant must be able to demonstrate an understanding of the study at his or her comprehension level and must have the ability to give verbal assent. If the legal guardian is court appointed, then the legal guardian must be able to provide documentation of court appointed guardianship.

Exclusion Criteria:

1. A diagnosis of ulcerative colitis or indeterminate colitis.
2. Requirement for immediate surgical, endoscopic or radiological intervention for perforation, sepsis, or intra-abdominal or perianal abscess.
3. History of colorectal cancer or dysplasia.
4. Positive stool test for Clostridium difficile via GDH/EIA two step testing method. PCR only testing will not be accepted. If patient is GDH positive and EIA negative, enrollment will be permitted.
5. Current medically significant infection.
6. Significant laboratory abnormalities;

   1. Hb < 7.0 g/dL, WBC < 2.5 x 103/mm3, Plt < 50 x 103/mm3.
   2. Creatinine ≥ 2x institutional ULN.
   3. Total bilirubin > 2.0 mg/dL, ALT > 2x institutional ULN. Elevated unconjugated bilirubin related to Gilbert's syndrome is allowed.
   4. Abnormal thyroid function tests.
7. Positive serology for HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV).
8. Positive screening test for tuberculosis (TB).
9. Treatment with any biologic medication within 4 weeks of first study drug dose (baseline) (see below section on washouts)
10. Received another IND within 5 half-lives of that agent baseline.
11. Malignancy within the last 5 years, excluding non-melanoma skin cancer.
12. Allergy to any component of the study drug.
13. Pregnant or lactating women.
14. Inability to comply with the study protocol or inability of the subject or the subject's legal guardian to provide informed consent.
15. Prior exposure to IL-2.
16. Uncontrolled cardiac angina or symptomatic congestive cardiac failure (NYHA Class III or IV).

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with serious and non-serious adverse events. | 8 weeks
  Enumeration of the serious and non-serious adverse events seen in the study. Enumeration of any dose limiting toxicity seen in the study.
Maximum effective dose | 8 weeks
  Identification of the dose cohort at which the MED occurs.

SECONDARY OUTCOMES:
Clinical Response | 8 weeks
  This is a composite endpoint. CDAI scores will be used to assess clinical activity. Moderate to severe CD, denoted by a CDAI score 220-450, is an inclusion criterion.
  Definition of Clinical Response. CDAI-100 response (≥100-point decrease in the CDAI score) at week 8 Composite Outcome: Clinical response and at least a 50% decrease in fecal calprotectin or CRP
Immunological Response | 12 weeks
  Enumeration of the number of subjects with a change in the absolute number of immune cells in the peripheral blood and lamina propria of subjects during the 8 weeks of treatment, and during the 4 weeks following cessation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Snapper, MD, PhD, Principal Investigator — Boston Children's Hospital; Jessica Allegretti, MD, MPH, Principal Investigator — Brigham and Women's Hosptial
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koreth J, Matsuoka K, Kim HT, McDonough SM, Bindra B, Alyea EP 3rd, Armand P, Cutler C, Ho VT, Treister NS, Bienfang DC, Prasad S, Tzachanis D, Joyce RM, Avigan DE, Antin JH, Ritz J, Soiffer RJ. Interleukin-2 and regulatory T cells in graft-versus-host disease. N Engl J Med. 2011 Dec 1;365(22):2055-66. doi: 10.1056/NEJMoa1108188. PMID 22129252
- [Background] Matsuoka K, Koreth J, Kim HT, Bascug G, McDonough S, Kawano Y, Murase K, Cutler C, Ho VT, Alyea EP, Armand P, Blazar BR, Antin JH, Soiffer RJ, Ritz J. Low-dose interleukin-2 therapy restores regulatory T cell homeostasis in patients with chronic graft-versus-host disease. Sci Transl Med. 2013 Apr 3;5(179):179ra43. doi: 10.1126/scitranslmed.3005265. PMID 23552371
- [Background] Saadoun D, Rosenzwajg M, Joly F, Six A, Carrat F, Thibault V, Sene D, Cacoub P, Klatzmann D. Regulatory T-cell responses to low-dose interleukin-2 in HCV-induced vasculitis. N Engl J Med. 2011 Dec 1;365(22):2067-77. doi: 10.1056/NEJMoa1105143. PMID 22129253
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095